Lead Principal Investigator: Dr. [Name], MD

Study title: A single arm, open label, multicenter study of the safety and efficacy of Nerivio for the acute

treatment of migraine in adolescents

#### RESEARCH PARTICIPANT INFORMATION AND CONSENT FORM

Site: Address:

**TITLE:** A single arm, open label, multicenter study of the safety

and efficacy of Nerivio for the acute treatment of migraine

in adolescents

PROTOCOL NO.: TCH004

(NCT04089761)

**SPONSOR:** Theranica Bioelectronics Ltd

**INVESTIGATOR:** XXXXXXXXXX

STUDY-RELATED PHONE NUMBER(S):

**Parents/Guardians:** You have the option of having your teen join this research study. This is a parental permission form. It explains this research study. If you decide that your teen can be in this study, you will sign this form to show that you agree. If you sign this form, you will receive a signed copy for your records.

**COMBINED Parental Permission/Assent:** If you are a parent or legal guardian of a teen who may take part in this study, permission from you is required. The assent (agreement) of your teen is also be required.

When we say "you" in this form, we mean you or your teen; "we" means the study doctor and other staff.

#### What is a research study?

- This consent form will explain the purpose, the procedures, the risks and possible benefits of taking part in this research study. Please review it carefully.
- The main goal of regular medical care is to help each patient. The main goal of a research study is to learn things to help future patients.
- We cannot promise that participation in this research study will help you.
- Your participation in this research study can result in side effects that are explained below.
- Someone from the research team will explain this study to you. Make sure all your questions are answered before you decide.
- Your participation in this study is voluntary. You may decide that your teen should not participate, and your teen may leave the study at any time.
- The quality of your teen's medical care will be the same whether he/she joins, declines, or decides to leave the study.

Lead Principal Investigator: Dr. [Name], MD

Study title: A single arm, open label, multicenter study of the safety and efficacy of Nerivio for the acute

treatment of migraine in adolescents

#### **Key information**

#### Reasons for the study

This research is being done to evaluate a new non-invasive drug-free acute treatment of migraine in adolescents aged 12-17 years old. You are being asked to take part in this study because your teen suffers from migraine.

The Nerivio device is indicated by the FDA for acute treatment of migraine with or without aura in patients 18 years of age or older who do not have chronic migraine. The purpose of this study is to assess the effect of the Nerivio device in the adolescence population. The Nerivio is a non-invasive neuromodulation device operated via a smartphone application. The device is worn on the upper arm, and the treatment is self-administered at the onset of a migraine attack. The device delivers non-painful electrical pulses to the skin that stimulate the body to initiate a pain inhibition mechanism in the brain. During the treatment, the users can adjust the intensity of the pulses according to how they tolerate it.

#### **Procedures**

In this study you will receive a device and you will be asked to treat your migraine attacks with it and report in the app the characteristics of the attacks at the beginning of the attack as well as at 2 and 24 hours after the attack has started. The study includes 4 visits to the clinic. We expect that you will be in this research study for 12 weeks after which you will have the option to continue in an 8-week free use phase with the device. More detailed information about the study procedures can be found under "detailed procedures".

#### Additional study information

The following is more detailed information about this study in addition to the key Information.

If I have questions or would like to know about:

| Who to talk to | You can call | At |
|---|---|---|
| <ul> <li>Emergencies</li> <li>General study questions</li> <li>Research-related injuries</li> <li>Any research concerns or complaints</li> </ul> | PI Name | Phone: xxx-xxx |
| <ul> <li>Emergencies</li> <li>General study questions</li> <li>Research-related injuries</li> <li>Any research concerns or complaints</li> </ul> | Lead Study Coordinator | Phone: xxx-xxx |
| Your child's rights as a research participant | Institutional Review Board This is a group of scientists and community members who make sure research meets legal and | Phone: 1-800-562-4789 or 360-252-2500. |

Lead Principal Investigator: Dr. [Name], MD

Study title: A single arm, open label, multicenter study of the safety and efficacy of Nerivio for the acute

treatment of migraine in adolescents

| Who to talk to | You can call | At |
|----------------|--------------------|----|
| | ethical standards. | |

## **Total number of participants**

We expect about 130 participants will be in this research study conducted in the USA and Israel, with up to 20 participants in this site.

## Who is doing the research study?

Dr. [Name] is in charge of this research study at [Site].

#### Who is funding the study?

This study is funded by Theranica. Theranica, the manufacturer of the Nerivio device being used in this study, provides the study device to the researcher or research participant without costs.

#### **Detailed procedures**

If you agree to be in the study, you will answer questions regarding your general medical state and your migraine in order to determine whether you are eligible to participate in the study. If you are a girl and have had your first period, we will ask you to supply a urine sample for pregnancy testing.

Each participant will receive a device to be used at home for the acute treatment of migraine attacks. The device produces electrostimulation parameters aimed to relief migraine pain. In addition, an app will be installed on your smartphone to control the device and record your migraine attacks and your feedback regarding the effect of the device on your migraine attacks.

The table below outlines what you will be responsible for during the course of this study.

| Schedule | What you do |
|---|---|
| Enrollment<br>Visit 1<br>(Day 0) | <ul> <li>Arrive to [Site], with one of your parents, for your scheduled appointment. Bring packages of any medications you are taking (for any medical condition).</li> <li>Eligibility assessment</li> <li>Meet with Dr. [Name], or one of the colleagues and/or the study team to answer questions about your general health and your migraine.</li> <li>If this form is received today, you and your parent(s) can take time to read it carefully and make sure all your questions and concerns are answered.</li> <li>You may request another appointment in case you would like to read this form at home and consult with family members or friends.</li> <li>If you are a girl and have had your first period, you will provide a urine sample for a pregnancy test.</li> </ul> |

Lead Principal Investigator: Dr. Namel, MD

Study title: A single arm, open label, multicenter study of the safety and efficacy of Nerivio for the acute

treatment of migraine in adolescents

| | <ul> <li>If you agree to participate, a member of the study staff will install the app on your smartphone. We will provide an explanation on how to operate the smartphone application.</li> <li>We will train you how to complete your migraine diary.</li> <li>.</li> </ul> |
|---|---|
| Run-in<br>phase<br>(Days 1-30) | <ul> <li>Complete the diary whenever you experience a migraine attack.</li> <li>Eligibility to continue in the study will be assessed based on your reports and compliance in the run-in phase.</li> <li>The study staff will contact you to schedule your next visit</li> </ul> |
| Device<br>training<br>Visit 2<br>(Day 31-37) | <ul> <li>You will receive a device.</li> <li>We will train you how to use the device and find the intensity level that is best for you</li> <li>You can ask us any questions.</li> <li>You will take the Nerivio home with you.</li> </ul> |
| Treatment phase Treatment of 4 migraine attacks, for up to 8 weeks | <ul> <li>Always have the device and your smartphone available.</li> <li>Use the device for the treatment of your migraine attacks at attack onset (and always with 60 minutes of onset).</li> <li>To comply, you: <ul> <li>Avoid taking rescue medication from the time of symptoms onset until 2 hours from treatment start (≈75 minutes from the end of the treatment).</li> <li>Report the 2-hour and the 24-hour post treatment feedback through the smartphone application</li> </ul> </li> <li>The application will ask you to rate your migraine pain level at the beginning of the treatment, after 2 hours, and after 24 hours post treatment on a scale of 0-3 (0= no pain; 1= mild; 2= moderate; 3= severe)</li> <li>Call the study team if there is any change in your medical condition.</li> <li>At the end of this phase, you will be contacted by a member of the study team to schedule your next visit.</li> </ul> |
| Free-use visit or Study exit (Visit 3) | <ul> <li>Arrive to [Site] for your scheduled appointment.</li> <li>Return the device.</li> <li>Meet with the study team to answer questions about your general health and your migraine.</li> <li>Indicate whether you are interested in the free-use extension phase. If you are interested, we will provide you a device for this extension phase during this visit. If you are not interested, this will be your end-of-study visit.</li> </ul> |
| Free-use<br>extension<br>phase (8<br>weeks) | <ul> <li>Treat all attacks as above, and report attack characteristics using the app at baseline, 2, and 24 hours post treatment, as above.</li> <li>At the end of this phase, you will be contacted by a research team member to schedule your end of study visit.</li> </ul> |
| End of study visit | <ul> <li>Arrive to [Site] for your scheduled appointment.</li> <li>Return the device.</li> </ul> |

Lead Principal Investigator: Dr. [Name], MD

Study title: A single arm, open label, multicenter study of the safety and efficacy of Nerivio for the acute

treatment of migraine in adolescents

#### Please note:

• The procedures above are crucial to the success of the study. If you feel that you will not be able to comply with these procedures, please reconsider your participation in the study and inform us about your hesitations.

• During the study, you may receive text messages or phone calls from the study team. The purpose of these is to follow-up on your progress in the study, check if you have any questions, and provide reminders regarding how to use the device. If you do not agree to receive occasional text messages and/or phone calls from the researchers, please notify the clinic staff before you sign this document.

## What are the risks and possible discomforts?

You may have side effects while participating in this study. The device used in this study may cause temporary mild side effects that should resolve shortly after the treatment. The side effects that were reported in previous studies include

- Warmth sensation
- Redness
- Numbness of the hand/arm
- Weakness of the arm
- Itching
- Tingling
- Muscle spasms

All the side effects were mild and resolved after the treatment without any need for medical interventions

You should talk to your study doctor about any side effects experienced while taking part in the study.

The Nerivio device was proven to be a safe technology, therefore the study is expected to have a minimal risk profile.

For more information about risks and side effects, ask your study doctor.

#### How will I find out about new information?

We will tell you about any new information that may affect your health, welfare or change your decision to be in this study.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## What are the possible benefits?

We cannot promise any benefits to you or others from your taking part in this research. However, you may experience relief in migraine pain and other symptoms without

Lead Principal Investigator: Dr. [Name], MD

Study title: A single arm, open label, multicenter study of the safety and efficacy of Nerivio for the acute

treatment of migraine in adolescents

having to take medications to treat your attacks in the course of the study. Furthermore, participating in this study may provide you the chance to receive up-to-date care, will help learn more on the effectiveness of the device for adolescents with migraine and it is hoped that this information will help in the treatment of future patients with conditions like yours.

Lastly, information gained from this research could lead Nerivio to help others with chronic migraine in the future.

# What are my alternatives? If I do not want to take part in the research study, are there other choices?

Participation in research is completely voluntary. Your decision to participate or not to participate will not affect the care you receive. Instead of being in this research study, your choices may include getting treatment or care for migraine without being in a study. Please talk to your doctor about your choices before deciding if you will take part in this study. Your alternatives include pain relieve medications and preventative treatments, physical therapy, nerve blocks, Botox, or the use of other nerve stimulators as well as not participating in this study or participating in another study to treat migraine headaches

#### Are there any additional costs?

You will not incur any additional costs by participating in this study. The study device will be provided at no charge to you by the study sponsor. You will not be charged for any study-related activities, including study visits.

#### Will I be paid?

If you agree to take part in this research study, we will pay you a total of \$200 for your time and effort in the form of a gift card. The compensation will be provided according to the completion of the study phases (see detailed procedures). After the run-in phase, you will receive \$50, after the treatment phase, you will receive \$100 and after the open label extension phase, you will receive additional \$50.

#### Change of mind/study withdrawal

You can leave the research at any time; it will not be held against you. If you decide to leave the research, contact the investigator so that the investigator can schedule a final visit and to discuss further care.

The person in charge of the research study or the sponsor can remove you from the research study without your approval. Possible reasons for removal include incompliance with the study protocol, concern about your safety, or early termination of the study.

#### **Privacy**

Efforts will be made to limit the use and disclosure of your personal information, including research study and medical records, to people who have a need to review this information. We cannot promise complete privacy. Organizations that may inspect and copy your information include the IRB and other representatives of this organization and

Lead Principal Investigator: Dr. [Name], MD

Study title: A single arm, open label, multicenter study of the safety and efficacy of Nerivio for the acute

treatment of migraine in adolescents

representatives from federal and state government oversight agencies such as the Food and Drug Administration. The sponsor, monitors, auditors, the IRB, the Food and Drug Administration will be granted direct access to your medical records to conduct and oversee the research. By signing this document, you are authorizing this access. We may publish the results of this research. However, we will keep your name and other identifying information confidential.

If you have questions about your privacy rights, please call the Western Institutional Review Board® (WIRB®) at 1-800-562-4789 or 360-252-2500.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Website will not include information that can identify you. At most, the Website will include a summary of the results. You can search this Website at any time.

## If injured in the study

If you believe that you have been injured as a result of this research, you should contact Dr. [Name] as soon as possible to discuss the concerns. The sponsor of the study has agreed to pay for reasonable and necessary expenses incurred by you for medical care. These expenses include any and all medical, hospitalization and hospitalization related expenses caused by the research procedures.

# <u>AUTHORIZATION TO USE AND DISCLOSE INFORMATION FOR</u> RESEARCH PURPOSES

To be in this research study you must also give your permission (or authorization) to use and disclose (or share) your "protected health information" (called PHI for short).

## What protected health information may be used and shared during this study?

Your health information that may be used for this study shared with others may include:

- Laboratory test results, diagnosis, and medications
- Written information, such as what is in your medical chart, or the record of your study visits
- Electronic information, which is information stored in computer systems.
- Verbal information, such as in phone calls made as part of this research study
- Information obtained during this research about
  - Past and present medical history
  - Diaries and questionnaires
  - Study procedures, treatments and follow-up
- Records about the study device

#### Who will share, receive and/or use your protected health information in this study?

- Staff at all the research study sites
- Personnel who provide services to you as part of this study

Lead Principal Investigator: Dr. [Name], MD

Study title: A single arm, open label, multicenter study of the safety and efficacy of Nerivio for the acute

treatment of migraine in adolescents

 Other individuals and organizations that need to use your PHI in connection with the research, including people at the sponsor and organizations that the sponsor may use to oversee or conduct the study.

- Representatives from federal and state government oversight agencies such as the Food and Drug Administration.
- Representatives from Western Institutional Review Board® (WIRB®), the group of people that oversee research at this institution.

If the researchers learn about potential serious harm to you or someone else or other public health concerns, it will be shared with the appropriate authorities.

## What if I decide not to give permission to use and share my health information?

By signing this consent form, you are giving permission to use and share your PHI. If you refuse to give permission, you will not be able participate in this research. You may choose to withdraw your permission at any time. A withdrawal of your permission to use and share your PHI would also include a withdrawal from participation in the research study.

## Will this permission expire?

Your permission will expire at the end of the study.

## Involvement of the General Practitioner (GP)/family doctor

With your consent, your GP will be informed of your involvement in the study. Any other medical practitioners who treat you (for example should you be admitted to the hospital for any reason) may also be informed.

#### Will your child's other medical care be impacted?

By signing this document, you / your child agree/s to participate in this research study and give permission to use and share you/your child's PHI for the purpose of this research study. If you refuse to sign this document, you/your child will not be able to participate in the study. However, you/your child's rights concerning treatment not related to this study, payment for services, enrollment in a health plan or eligibility of benefits will not be affected.

Lead Principal Investigator: Dr. [Name], MD

Study title: A single arm, open label, multicenter study of the safety and efficacy of Nerivio for the acute

treatment of migraine in adolescents

## **SIGNATURES**

The research team has discussed this study with you and answered all your questions. Like any research, the researchers cannot predict exactly what will happen. Once you have had enough time to consider whether you/your child should participate in this research, you will document your permission by signature below.

| You will receive a copy of the | nis signed docum | ent for your records. | |
|---|---|---|---|
| Printed Name of Research Pa | articipant | _ | |
| Street: | | | |
| City: | State: | Zip: | |
| Signature of Parent or Legall Representative* | y Authorized | Date | |
| * If signed by a legally authority must be provided | orized representat | ive, a description of such re | <del></del> epresentative's |
| Name of Person Conducting<br>Informed Consent Discussion | | Role in the study | |
| Signature | | <br>Date | |